CLINICAL TRIAL: NCT03999333
Title: A Prospective Pilot Study to Evaluate the Effect of Virtual Reality As a Treatment Option for Pain in Patients with Functional Pancreaticobiliary Disorder or Type 3 Sphincter of Oddi Dysfunction
Brief Title: Virtual Reality in SOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Simon K. Lo, M.D., Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00057560
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Sphincter of Oddi Dysfunction
MeSH Terms: conditions — Sphincter of Oddi Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Virtual Reality (Experimental): Every participant is provided with a VR headset
  Interventions: Device: Virtual Reality (Oculus Go)

INTERVENTIONS:
Device: Virtual Reality (Oculus Go) — Participants will self-administer virtual reality intervention, in addition to standard of care treatment for pain. There will be 6 weeks of weeks of monitoring period (2 weeks before, 4 weeks during, and 2 weeks after the virtual reality intervention).

SUMMARY:
Patients with classic type-3 Sphincter of Oddi dysfunction have chronic debilitating pain not amenable to pharmacologic or endoscopic therapy. Previous studies have shown benefits of virtual reality (VR) for pain management through immersive three-dimensional (3D) multisensory experiences, but only in short-term inpatient settings.

The impact of VR for chronic pain in patients with SOD III in an outpatient setting is being evaluated in this pilot study.

DETAILED DESCRIPTION:
The pain management for type-3 Sphincter of Oddi dysfunction remains a significant clinical challenge and the current therapeutic outcome is often frustrating and may lead to addiction of opioid pain medication. Virtual reality (VR) has emerged as a viable option for pain management, but its usage has been limited to short-term inpatient clinical trials or experimental settings. In the proposed study, we will determine the long-term efficacy of VR intervention on pain management in patients with SOD type 3.

The study involves an initial screening visit and one follow-up visit at the end of the 6-week study.

The participants will receive self administered VR intervention, in additional to standard-of-care treatment for pain. The study also includes 6 weeks of monitoring period (2 weeks before, 4 weeks during, and 2 weeks after the VR intervention).

If the aims of the research are achieved, the study will demonstrate that virtual reality intervention may be used as a new method for pain management. This may lead to reduction in usage of opioid pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic biliary type abdominal pain (RUQ pain, pain radiates to the right flank, scapula, or shoulder, or pain that stimulates gallbladder symptoms)
* Pancreatic pain (epigastric or left upper quadrant pain, pain that is exacerbated by some food, or pain that radiates to the back) for at least 3 months prior to the study
* absence of abnormal liver and pancreas chemistry or abnormal abdominal imaging
* average pain score of greater than or equal to 3 out of 10 on the numeric rating scale (NRS) for at least the average of 3 episodes each week
* Subjects on antidepressants for pain control should take the medication for a minimum of one month prior to the baseline assessment.
* Patients with SOD with depressive and/or anxiety disorders who receive psychopharmacologic treatment must be on stable medication dose for at least 6 weeks.
* Patients with access to a cell phone, able to speak, read, and write English will be enrolled.

Exclusion Criteria:

* Patients with evidence for acute or chronic pancreatitis, biliary stones, or bile duct strictures.
* Patients who have had prior sphincterotomy must have had the procedure at 3 months prior to the start of the study.
* Patients with a history of motion sickness and vertigo and anyone experiencing active nausea or vomiting (including pregnant women) will be excluded.
* Patients with a history of seizures or epilepsy will also be excluded to limit the theoretical risk of inducing seizures with VR.
* Presence of significant psychiatric disorders or any conditions that, in the investigator's opinion make the subject unsuitable for study participation will be reason for exclusion.
* Non-English speaking subjects or subjects unable to consent to study due to cognitive difficulty will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Pain scores | 6 weeks
  Pain scores will be measured using the Numeric Rating Scale (NRS) for at least 3 episodes each week. The NRS measures pain on a scale of 0 to 10, with 0 signifying no pain and 10 signifying the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lo, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No